CLINICAL TRIAL: NCT01883323
Title: Phase II Study Evaluating The Infusion Of Autologous Tumor-Infiltrating Lymphocytes (TILs) And Low-Dose Interleukin-2 (IL-2) Therapy Following A Preparative Regimen Of Non-Myeloablative Lymphodepletion Using Cyclophosphamide And Fludarabine In Patients With Metastatic Melanoma
Brief Title: Tumor-Infiltrating Lymphocytes And Low-Dose Interleukin-2 Therapy Following Cyclophosphamide And Fludarabine In Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILs-002-MEL
Record Dates: First submitted 2013-06-11; First posted 2013-06-21 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Metastatic, Stage III or Stage IV, Melanoma
Keywords: Measurable; Unresectable; Stage III; Stage IV; Metastatic; Melanoma; Tumor-Infiltrating Lymphocytes; Low-Dose Interleukin-2; Cyclophosphamide; Fludarabine
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukins; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide and Fludarabine followed by TILs and IL-2 (Experimental): Cyclophosphamide, i.v., 60mg/kg per day for 2 days and Fludarabine, i.v., 25mg/m2 per day for 5 days; then Tumor-Infiltrating Lymphocytes, i.v., 1x10^10 - 1.6x10^11 cells and Low-Dose Interleukin, i.v., 125,000 IU/kg subcut per day, for 2 weeks (2 days rest between each week)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor-Infiltrating Lymphocytes; Biological: Low-Dose Interleukin

INTERVENTIONS:
Drug: Cyclophosphamide — i.v., 60mg/kg per day for 2 days
  Other Names: CYTOXAN, PROCYTOX
Drug: Fludarabine — i.v., 25mg/m2 per day for 5 days
  Other Names: FLUDARA
Biological: Tumor-Infiltrating Lymphocytes — i.v., 1x10^10 - 1.6x10^11 cells
Biological: Low-Dose Interleukin — i.v., 125,000 IU/kg subcut per day, for 2 weeks (2 days rest between each week)
  Other Names: Aldesleukin, Proleukin, Recombinant Human Interleukin 2

SUMMARY:
This is a phase II clinical study for patients with metastatic (the cancer has spread to other parts of the body) melanoma. Patients will receive an infusion (given by vein) of autologous tumor infiltrating lymphocytes (TILs). TILs are a type of white blood cells that recognizes tumor cells and enter them which causes the tumor cells to break down.

Prior to the cell infusion, patients will receive a two drugs cyclophosphamide and fludarabine to prepare the body to receive the TILs. After cell infusion, patients will receive low-dose interleukin-2 therapy which is an approved drug to treat melanoma. This study will see how useful this regimen is in treating metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria (Eligibility for TIL Evaluation):

* Must have measurable, unresectable stage III or stage IV melanoma
* Suitable tumor for collection
* If tumor is suitable for collection, patient must be suitable for surgery
* Patient must be 18 years of age or older
* Performance status of ECOG 0 or 1
* Life expectancy > 5 months from date of consent of TIL evaluation
* Willing to be tested for transmissible diseases
* For patients with a history of allergy to penicillin, gentamycin, streptomycin, or anti-fungals, the ability to generate TILs will be confirmed with the cell manufacturing laboratory

Inclusion Criteria (Eligibility for Treatment):

* Signed and dated the informed consent
* No brain metastases or stable brain metastases for 3 months following definitive treatment.
* Life expectancy > 3 months from the date of consent for TILs treatment
* TILs are suitable for use as determined by laboratory
* More than 30 days since any prior systemic therapy at the time of the cell infusion, or more than six weeks since prior nitrosurea therapy. For patients with prior ipilimumab therapy, at least six weeks must elapse between the last ipilimumab dose and the start of study treatment. All side effects from previous treatment must have recovered to an acceptable grade level.
* Adequate organ function
* Must have positive EBV titres
* Women of child-bearing potential must have a negative pregnancy test. Patients of both genders must be willing to practice birth control during treatment and for 6 months post completion of IL-2 treatment.

Exclusion Criteria:

* Requiring systemic steroid therapy
* HIV positive
* With active hepatitis B or hepatitis C, syphilis, or HTLV
* Must not have any active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, uncontrolled psychiatric disorders, or other conditions that may affect following study procedures.
* Have no active underlying cardiac illnesses defined by positive stress test, LVEF<40% or ongoing life-threatening arrhythmias
* Abnormal lung function test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Clinical response to treatment | 6 weeks after treatment

SECONDARY OUTCOMES:
Number occurrences and severity of side effects | Starting at first dose of study treatment up to 10 years
Number of patients with an immunity and no immunity to the study treatment | From start of study up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Butler Marcus, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nguyen LT, Saibil SD, Sotov V, Le MX, Khoja L, Ghazarian D, Bonilla L, Majeed H, Hogg D, Joshua AM, Crump M, Franke N, Spreafico A, Hansen A, Al-Habeeb A, Leong W, Easson A, Reedijk M, Goldstein DP, McCready D, Yasufuku K, Waddell T, Cypel M, Pierre A, Zhang B, Boross-Harmer S, Cipollone J, Nelles M, Scheid E, Fyrsta M, Lo CS, Nie J, Yam JY, Yen PH, Gray D, Motta V, Elford AR, DeLuca S, Wang L, Effendi S, Ellenchery R, Hirano N, Ohashi PS, Butler MO. Phase II clinical trial of adoptive cell therapy for patients with metastatic melanoma with autologous tumor-infiltrating lymphocytes and low-dose interleukin-2. Cancer Immunol Immunother. 2019 May;68(5):773-785. doi: 10.1007/s00262-019-02307-x. Epub 2019 Feb 11. PMID 30747243